CLINICAL TRIAL: NCT06839326
Title: Comparison of the Effectiveness of Autologous Conditioned Serum and Platelet-rich Plasma in Temporomandibular Joint Osteoarthritis; A Randomized Prospective Study
Brief Title: Efficacy of Autologous Conditioned Serum in Temporomandibular Joint Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Rojdan Ferman GÜNEŞ UYSAL, Assistant professor, Batman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BatmanU-DF-RFGU-02
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Joint Osteoarthritis
Keywords: Arthrocentesis, TMJ; Platelet-Rich Plasma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and the second physician who performed post-operative control measurements, will be unaware of the treatment given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Autologous Conditioned Serum (Experimental): Approximately 10 mL of venous blood will be drawn from patients receiving Autologous Conditioned Serum (ACS) treatment and placed into a specialized tube (Genesis Biomedical, Sanakin®-ACRS kit) containing glass beads designed to facilitate the adhesion of monocytes and other sticky molecules. The tube will then be incubated at 37°C for 3 hours, following the manufacturer's instructions.
  After the incubation period, the tube will be centrifuged at 4000 rpm for 5 minutes. The resulting serum will then be transferred into a new syringe for intra-articular injection. After completing the arthrocentesis, the needle in the second entry point will be removed, and 1 mL of ACS will be injected into the joint.
  Interventions: Biological: Autologous Conditioned Serum, Genesis Biyomedikal, Sanakin®-Acrs produce
- Group 2 Platelet Rich Plasma (Active Comparator): For patients receiving platelet rich plasma (PRP) treatment, approximately 10 mL of venous blood will be collected in a tube containing sodium citrate and centrifuged at 3000 rpm for 10 minutes.
  After centrifugation, the buffy coat (the middle layer) and a portion of the upper plasma layer will be aspirated into a syringe, excluding the lower layer rich in erythrocytes.
  After completing the arthrocentesis, the needle in the second entry point will be removed, and 1 mL of PRP will be injected into the joint.
  Interventions: Biological: Platelet Rich Plasma
- Group 3 Only Arthrocentesis (Placebo Comparator): Arthrocentesis Procedure: Arthrocentesis and intra-articular injection will be performed under sterile conditions. Before the procedure, the skin of the ear and preauricular region will be cleansed with povidone-iodine, and the surrounding areas will be covered with a sterile drape. The joint area will then be anesthetized with approximately 1 cc of lidocaine (Jetokain®; Adeka).The injection entry points will be determined along the tragus-lateral canthus line. The first entry point located 10 mm anterior and 2 mm inferior to the tragus. The second entry point located 20 mm anterior and 8 mm inferior to the tragus. With the patient's mouth open, a 20-gauge needle will be inserted through the designated entry points, and irrigation with approximately 150 mL of 5% Ringer's lactate solution will be performed.
  Interventions: Other: Control Group/ Only Arthrocentesis

INTERVENTIONS:
Biological: Autologous Conditioned Serum, Genesis Biyomedikal, Sanakin®-Acrs produce — Arthrocentesis and 1ml ACS injection will be performed twice in total, two weeks apart.
  Arms: Group 1 Autologous Conditioned Serum
Biological: Platelet Rich Plasma — Arthrocentesis and 1ml PRP injection will be performed twice in total, two weeks apart.
  Arms: Group 2 Platelet Rich Plasma
Other: Control Group/ Only Arthrocentesis — Arthrocentesis will be performed twice in total, two weeks apart.
  Arms: Group 3 Only Arthrocentesis

SUMMARY:
Temporomandibular joint (TMJ) disorders are health conditions that can occur at any age and are recognized as the most common cause of chronic pain, affecting 5-12% of the population. Pain in the TMJ region can lead to limitations in mouth opening and lateral movements of the mandible.

In cases where conservative treatments are insufficient for TMJ disorders and osteoarthritis, symptoms can be alleviated through arthrocentesis, a minimally invasive procedure with a low risk of complications, or through various intra-articular injection applications following arthrocentesis.

This study aims to compare the clinical efficacy of intra-articular applications of platelet-rich plasma (PRP) and autologous conditioned serum (ACS), both derived from the patient's own blood, in order to evaluate their impact on treatment outcomes and their potential role in enhancing patient care in routine clinical practice."

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) disorders are health conditions that can occur at any age and negatively impact quality of life. One of the treatment methods for this condition includes arthrocentesis and intra-articular injections.

Among the cytokines identified in orthopedic and trauma-related diseases, interleukin-1 (IL-1) has been shown to have particular significance. Increased local cytokine release triggers the destruction of hyaline cartilage and matrix, leading to osteoarthritis and worsening symptoms. Although the details vary, published studies suggest that when IL-1Ra is present at concentrations 10 to 10,000 times higher than IL-1, all IL-1 receptors and IL-1-triggered reactions can be effectively blocked.

With the Sanakin®-ACRS kit developed by Genesis Biomedical, a patient's blood is drawn, incubated, and then centrifuged, resulting in a serum rich in IL-1Ra and growth factors-known as autologous conditioned serum (ACS). Studies have demonstrated that ACS injections yield highly successful results in treating knee and TMJ osteoarthritis. Additionally, numerous studies have shown that platelet-rich plasma (PRP), which contains a high concentration of growth factors, is also highly effective in wound healing.

This study is designed to compare the effectiveness of PRP and ACS injections-both derived from the patient's own blood but prepared using different methods-in alleviating symptoms associated with temporomandibular joint (TMJ) disorders. The investigation aims to assess their efficacy as accessible, cost-effective, and low-risk treatment alternatives."

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Previously received conservative treatment but no improvement in symptoms
* Patients with TMJ osteoarthritis

Exclusion Criteria:

* Patients who have experienced TMJ trauma or have undergone surgical procedures in this region will be excluded from the study.
* Patients with facial growth disorders, systemic inflammatory joint diseases, condylar pathologies, or signs of myalgia
* Patients who are pregnant or in the lactation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain level | Measurements will be conducted preoperatively, as well as at 1 week, 1 month, 3 months, and 6 months postoperatively
  All patients' initial and post-operative pain levels will be measured with a 10-unit Visual Analogue Scale (VAS).
Maximum mouth opening measurement | Measurements will be conducted preoperatively, as well as at 1 week, 1 month, 3 months, and 6 months postoperatively
  The maximum mouth opening and the amount of lateral and protrusive movement of the mandible will be noted in millimeters with the help of a caliper

CONTACTS AND LOCATIONS:
Overall Officials: Rojdan F GÜNEŞ UYSAL, PhD, Principal Investigator — Batman University; İbrahim UYSAL, PhD, Study Chair — Dicle University
Locations (1):
- Batman University, Batman, Centre/Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No